CLINICAL TRIAL: NCT06380114
Title: Stand Up 2 HPV: Standing Orders to Improve HPV Vaccination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Cynthia Rand, Professor, Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00009296; R01CA270276 (NIH)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-03

CONDITIONS: Hpv
MeSH Terms: conditions — Papillomavirus Infections | interventions — Standing Orders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Communication Training (Active Comparator): Practice personnel (providers and nurses) receive training in communication about HPV vaccination.
  Interventions: Behavioral: Communication
- Communication Training + Standing Orders Training/Implementation (Experimental): Practice personnel (providers and nurses) receive training in communication about HPV vaccination and training in the implementation of standing orders for HPV vaccination.
  Interventions: Behavioral: Communication; Behavioral: Standing Orders

INTERVENTIONS:
Behavioral: Communication — Practice personnel (providers and nurses) receive training in communication about HPV vaccination via an online learning module.
Behavioral: Standing Orders — Practice personnel (providers and nurses) receive training in the implementation of standing orders for HPV vaccination via an online learning module and meetings with the study team.
  Arms: Communication Training + Standing Orders Training/Implementation

SUMMARY:
Each year in the U.S., ≥20,000 women and 14,000 men are affected by HPV-related cancers, including cervical and oropharyngeal cancer. However, in 2020, only 59% of U.S. adolescents aged 13-17 were up-to-date for HPV vaccination, and rates for 11-12 year olds, the primary target age group for HPV vaccination (when the immune reaction is better and before exposure to HPV infection), are even lower. Standing orders (written protocols that authorize designated members of the healthcare team to vaccinate without first obtaining a patient-specific physician order) have been shown to work in inpatient settings and for adults, but have not been evaluated for HPV vaccine, which some parents consider controversial. Also, the ways in which organizational readiness for change (resources, motivation, staff attributes, leadership support and culture) moderate the effect of standing orders has not been studied. A physician's recommendation is correlated with HPV vaccine acceptance, and the investigators have developed a successful online, interactive, communication education program that will be adapted to train nurses and staff in addition to physicians. The investigators propose testing standing orders for HPV vaccine in an Accountable Care Organization (ACO) in Western New York, and assessing which provider and practice factors moderate the effect of standing orders. Advantages of this setting include a diverse group of rural, urban and suburban practices, and the ACO provides data infrastructure and analytics that allow practices to evaluate vaccination rates in real time.

Using a 2-arm cluster randomized trial (n=40 practices), the investigators will assess the effectiveness of standing orders (SO) + HPV communication education (intervention arm) relative to HPV communication education alone (control arm) on HPV vaccination for 9-17 year-olds.

ELIGIBILITY:
Inclusion Criteria:

* active patient in AHP practice

Exclusion Criteria:

* patient belonging to a practice with >80% UTD baseline HPV vaccination rate for ages 13-17
* patient belonging to a practice with <20 11-12 year-olds eligible for an HPV dose

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16000 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Patient-Level Captured Opportunities for HPV Vaccination | 12-month baseline compared to 12-month intervention compared to 12-month maintenance (control arm vs intervention arm)
  The percentage of HPV vaccine eligible patients, aged 9-17, with a practice visit during the specified timeframe of interest who receive >=1 HPV vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center (URMC), Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with investigators upon request as part of a collaboration.